CLINICAL TRIAL: NCT02681302
Title: Phase Ib-IIA Study of Combined Check Point Inhibition After Autologous Hematopoietic Stem Cell Transplantation in Patients at High Risk for Post-transplant Recurrence
Brief Title: Check Point Inhibition After Autologous Stem Cell Transplantation in Patients at High Risk of Post Transplant Recurrence
Acronym: CPIT001
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of Accrual
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0048
Record Dates: First submitted 2016-01-29; First posted 2016-02-12 (Estimated); Results first posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma; Lymphoma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Participants (Experimental): * Ipilimumab 1 mg/kg; 6 doses Weeks 1, 4, 7, 10, 16, 22
  * Nivolumab 3 mg/kg; 12 doses Weeks 1, 4, 7, 10, 12, 14, 16, 18, 20, 22, 24, 26
  Interventions: Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Ipilimumab — 1 mg/kg; 6 doses Weeks 1, 4, 7, 10, 16, 22
  Other Names: Yervoy
Drug: Nivolumab — 3 mg/kg; 12 doses Weeks 1, 4, 7, 10, 12, 14, 16, 18, 20, 22, 24, 26
  Other Names: Opdivo

SUMMARY:
The goal of this study is to determine the safety and clinical effect of combined checkpoint inhibition administered after autologous hematopoietic stem cell transplantation in each of six clinical cohorts of high risk and recurrent disease. In addition to assessing the incidence and severity of adverse events and rates of complete response and progression free survival, investigators intend to monitor immune reconstitution, phenotype and TCR repertoire throughout treatment and at the time of disease progression. Investigators will also analyze the gut microbiome prior to conditioning, throughout treatment, post-transplant and at time of relapse.

DETAILED DESCRIPTION:
This is a phase Ib-IIA study of post-transplant combined check point inhibitors for patients with a high risk of relapse (>50%) after an autologous hematopoietic stem cell transplant.

Patients will accrue to study by disease groups and followed separately by group for incidence and severity of toxicity, ability to receive intended schedule of combined check point inhibitors and for complete response and progression free survival (PFS) rates. Complete response and progression free survival rates will be compared to published standards for each disease group. Expected PFS at 18 months for all post-transplant groups without check point inhibitors is less than 50%. Each group with PFS at 18 months in 4 or more patients (57%) will be considered for eligibility in a successor phase IIB expansion trial.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signed and dated IRB/IEC approved written informed consent form in accordance with regulatory and local guidelines.
2. Be 18 years or older and 80 years or younger on the day of signing consent
3. Have a confirmed diagnosis of:

   * (GROUP A) De novo diffuse large B cell lymphoma that fails to achieve a PET negative complete response to primary rituximab and anthracycline based multi-agent chemotherapy and at least maintains stable disease after salvage chemotherapy or present double/triple hit features defined by overexpression by standard immunohistochemistry of c-MYC plus BCL2 and/or BCL6 or presence of chromosomal translocations as detected by break-apart FISH involving IGH/MYC plus IGH/BCL2 and/or IGH/BCL6 and who only received standard chemoimmunotherapy with rituximab, cyclophosphamide, vincristine and prednisone (R-CHOP) for induction and present at least stable disease after consolidation or salvage chemotherapy. Stable disease (SD) for lymphoma is defined in Appendix B: Lugano Classification for Response Assessment of Non-Hodgkin Lymphoma.
   * (GROUP B) Recurrent high-risk diffuse large B cell lymphoma defined as relapsing within one year of completion of rituximab and anthracycline based multi-agent chemotherapy or a sAAIPI (second-line age-adjusted International Prognostic Index) intermediate or high at relapse or acquisition of double/triple hit features upon relapse (as defined in group A) and at least stable disease after salvage chemotherapy. Patients with an initial diagnosis of low-grade/indolent non-Hodgkin lymphoma (i.e. follicular, marginal zone) who present relapse with histologic transformation to diffuse large B cell lymphoma (confirmed by biopsy) and meet the definition for high-risk as presented above, are also eligible.
   * (GROUP C) De novo high-risk T cell lymphoma with at least stable disease after primary therapy. High risk T cell lymphoma is defined as Stage III or IV disease at presentation and/or failure to achieve CR after frontline chemotherapy. Patients with ALK-positive ALCL will be excluded from the trial. Patients with ALK-negative ALCL in complete response will be excluded from the trial.
   * (GROUP D) Recurrent T cell lymphoma with at least stable disease after salvage therapy. Patients with ALK-positive ALCL will be excluded from the trial.
4. Be deemed eligible for an autologous stem cell transplantation according to the institutional guidelines of the Blood and Marrow Transplantation Program at John Theurer Cancer Center at Hackensack University Medical Center
5. Have an ECOG performance status of 2 or lower
6. Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug.
7. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Female subjects of childbearing potential should agree to ongoing pregnancy testing, to be performed prior to each dosing of ipilimumab and nivolumab. See Note below for definition of WOCBP.
8. Women must not be breastfeeding.
9. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab, and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product, even if they have had a vasectomy. Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception). See Note below for definition of WOCBP.
10. Females of childbearing potential must be willing to use two methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 2 years. See Note below for definition of WOCBP.
11. Allowable transplant preparative regimens are the following:

    * For non-Hodgkin lymphoma groups (A, B,C,D) BEAM: carmustine 300 mg/m2 day -6, etoposide 200 mg/m2 and cytarabine 200 mg/m2 days -5 to -2, melphalan 140 mg/m2 day -1
    * For Myeloma groups (E and F) Melphalan 200 mg/m2 day -1

Exclusion Criteria:

1. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability. Note: Subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if > 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
2. Is unable or unwilling to sign informed consent.
3. Has an active, known, or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
4. Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Note: Subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if > 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
5. As there is potential for hepatic toxicity with nivolumab or nivolumab/ipilimumab combinations, drugs with a predisposition to hepatoxicity should be used with caution in patients treated with nivolumab-containing regimen.
6. Has received an allogeneic stem cell transplant.
7. Has a history of hypersensitivity to nivolumab, ipilimumab, or any of its excipients, or severe hypersensitivity reaction to any previous monoclonal antibody.
8. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to Day 1 of checkpoint inhibitor treatment administration or who has not recovered (i.e., t administration mAb) within 4 weeks prior to dose of trial treatment. Rituximab within that period is allowed.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Note: Subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if > 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Has an active infection requiring intravenous systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 23 weeks for females and 31 weeks for males after the last dose of trial treatment.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2 agent, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways.
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) or known acquired immunodeficiency syndrome (AIDS).
17. Has positive test for Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected) indicating acute or chronic infection, as tested for transplant.
18. Has received a live vaccine within 30 days of planned start of study therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Donato, MD, Principal Investigator — Hackensack Meridian Health
Locations (2):
- United States (2):
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Hackensack University medical Center, Hackensack, New Jersey

REFERENCES:
- [Background] Philip T, Guglielmi C, Hagenbeek A, Somers R, Van der Lelie H, Bron D, Sonneveld P, Gisselbrecht C, Cahn JY, Harousseau JL, et al. Autologous bone marrow transplantation as compared with salvage chemotherapy in relapses of chemotherapy-sensitive non-Hodgkin's lymphoma. N Engl J Med. 1995 Dec 7;333(23):1540-5. doi: 10.1056/NEJM199512073332305. PMID 7477169
- [Background] Gisselbrecht C, Glass B, Mounier N, Singh Gill D, Linch DC, Trneny M, Bosly A, Ketterer N, Shpilberg O, Hagberg H, Ma D, Briere J, Moskowitz CH, Schmitz N. Salvage regimens with autologous transplantation for relapsed large B-cell lymphoma in the rituximab era. J Clin Oncol. 2010 Sep 20;28(27):4184-90. doi: 10.1200/JCO.2010.28.1618. Epub 2010 Jul 26. PMID 20660832
- [Background] Kumar SK, Lee JH, Lahuerta JJ, Morgan G, Richardson PG, Crowley J, Haessler J, Feather J, Hoering A, Moreau P, LeLeu X, Hulin C, Klein SK, Sonneveld P, Siegel D, Blade J, Goldschmidt H, Jagannath S, Miguel JS, Orlowski R, Palumbo A, Sezer O, Rajkumar SV, Durie BG; International Myeloma Working Group. Risk of progression and survival in multiple myeloma relapsing after therapy with IMiDs and bortezomib: a multicenter international myeloma working group study. Leukemia. 2012 Jan;26(1):149-57. doi: 10.1038/leu.2011.196. Epub 2011 Jul 29. PMID 21799510
- [Background] Rezvani AR, Kanate AS, Efron B, Chhabra S, Kohrt HE, Shizuru JA, Laport GG, Miklos DB, Benjamin JE, Johnston LJ, Arai S, Weng WK, Negrin RS, Strober S, Lowsky R. Allogeneic hematopoietic cell transplantation after failed autologous transplant for lymphoma using TLI and anti-thymocyte globulin conditioning. Bone Marrow Transplant. 2015 Oct;50(10):1286-92. doi: 10.1038/bmt.2015.149. Epub 2015 Jul 6. PMID 26146806
- [Background] Donato ML, Siegel DS, Vesole DH, McKiernan P, Nyirenda T, Pecora AL, Baker M, Goldberg SL, Mato A, Goy A, Rowley SD. The graft-versus-myeloma effect: chronic graft-versus-host disease but not acute graft-versus-host disease prolongs survival in patients with multiple myeloma receiving allogeneic transplantation. Biol Blood Marrow Transplant. 2014 Aug;20(8):1211-6. doi: 10.1016/j.bbmt.2014.04.027. Epub 2014 May 2. PMID 24792872
- [Background] Armand P, Nagler A, Weller EA, Devine SM, Avigan DE, Chen YB, Kaminski MS, Holland HK, Winter JN, Mason JR, Fay JW, Rizzieri DA, Hosing CM, Ball ED, Uberti JP, Lazarus HM, Mapara MY, Gregory SA, Timmerman JM, Andorsky D, Or R, Waller EK, Rotem-Yehudar R, Gordon LI. Disabling immune tolerance by programmed death-1 blockade with pidilizumab after autologous hematopoietic stem-cell transplantation for diffuse large B-cell lymphoma: results of an international phase II trial. J Clin Oncol. 2013 Nov 20;31(33):4199-206. doi: 10.1200/JCO.2012.48.3685. Epub 2013 Oct 14. PMID 24127452
- [Background] Ansell SM, Lesokhin AM, Borrello I, Halwani A, Scott EC, Gutierrez M, Schuster SJ, Millenson MM, Cattry D, Freeman GJ, Rodig SJ, Chapuy B, Ligon AH, Zhu L, Grosso JF, Kim SY, Timmerman JM, Shipp MA, Armand P. PD-1 blockade with nivolumab in relapsed or refractory Hodgkin's lymphoma. N Engl J Med. 2015 Jan 22;372(4):311-9. doi: 10.1056/NEJMoa1411087. Epub 2014 Dec 6. PMID 25482239
- [Background] Weber J. Immune checkpoint proteins: a new therapeutic paradigm for cancer--preclinical background: CTLA-4 and PD-1 blockade. Semin Oncol. 2010 Oct;37(5):430-9. doi: 10.1053/j.seminoncol.2010.09.005. PMID 21074057
- [Background] O'Day SJ, Hamid O, Urba WJ. Targeting cytotoxic T-lymphocyte antigen-4 (CTLA-4): a novel strategy for the treatment of melanoma and other malignancies. Cancer. 2007 Dec 15;110(12):2614-27. doi: 10.1002/cncr.23086. PMID 18000991
- [Background] Larkin J, Chiarion-Sileni V, Gonzalez R, Grob JJ, Cowey CL, Lao CD, Schadendorf D, Dummer R, Smylie M, Rutkowski P, Ferrucci PF, Hill A, Wagstaff J, Carlino MS, Haanen JB, Maio M, Marquez-Rodas I, McArthur GA, Ascierto PA, Long GV, Callahan MK, Postow MA, Grossmann K, Sznol M, Dreno B, Bastholt L, Yang A, Rollin LM, Horak C, Hodi FS, Wolchok JD. Combined Nivolumab and Ipilimumab or Monotherapy in Untreated Melanoma. N Engl J Med. 2015 Jul 2;373(1):23-34. doi: 10.1056/NEJMoa1504030. Epub 2015 May 31. PMID 26027431
- [Background] Fong L, Small EJ. Anti-cytotoxic T-lymphocyte antigen-4 antibody: the first in an emerging class of immunomodulatory antibodies for cancer treatment. J Clin Oncol. 2008 Nov 10;26(32):5275-83. doi: 10.1200/JCO.2008.17.8954. Epub 2008 Oct 6. PMID 18838703
- [Background] Postow MA, Chesney J, Pavlick AC, Robert C, Grossmann K, McDermott D, Linette GP, Meyer N, Giguere JK, Agarwala SS, Shaheen M, Ernstoff MS, Minor D, Salama AK, Taylor M, Ott PA, Rollin LM, Horak C, Gagnier P, Wolchok JD, Hodi FS. Nivolumab and ipilimumab versus ipilimumab in untreated melanoma. N Engl J Med. 2015 May 21;372(21):2006-17. doi: 10.1056/NEJMoa1414428. Epub 2015 Apr 20. PMID 25891304
- [Background] Sledzinska A, Menger L, Bergerhoff K, Peggs KS, Quezada SA. Negative immune checkpoints on T lymphocytes and their relevance to cancer immunotherapy. Mol Oncol. 2015 Dec;9(10):1936-65. doi: 10.1016/j.molonc.2015.10.008. Epub 2015 Oct 26. PMID 26578451
- [Background] Antonia SJ, Bendell JC, Taylor MH. Phase I/II study of nivolumab with or without ipilimumab for treatment of recurrent small cell lung cancer (SCLC): CA209-032. ASCO Annual Meeting. 2015.
- [Background] Taur Y, Jenq RR, Ubeda C, van den Brink M, Pamer EG. Role of intestinal microbiota in transplantation outcomes. Best Pract Res Clin Haematol. 2015 Jun-Sep;28(2-3):155-61. doi: 10.1016/j.beha.2015.10.013. Epub 2015 Oct 22. PMID 26590773
- [Background] Iida N, Dzutsev A, Stewart CA, Smith L, Bouladoux N, Weingarten RA, Molina DA, Salcedo R, Back T, Cramer S, Dai RM, Kiu H, Cardone M, Naik S, Patri AK, Wang E, Marincola FM, Frank KM, Belkaid Y, Trinchieri G, Goldszmid RS. Commensal bacteria control cancer response to therapy by modulating the tumor microenvironment. Science. 2013 Nov 22;342(6161):967-70. doi: 10.1126/science.1240527. PMID 24264989
- [Background] Viaud S, Saccheri F, Mignot G, Yamazaki T, Daillere R, Hannani D, Enot DP, Pfirschke C, Engblom C, Pittet MJ, Schlitzer A, Ginhoux F, Apetoh L, Chachaty E, Woerther PL, Eberl G, Berard M, Ecobichon C, Clermont D, Bizet C, Gaboriau-Routhiau V, Cerf-Bensussan N, Opolon P, Yessaad N, Vivier E, Ryffel B, Elson CO, Dore J, Kroemer G, Lepage P, Boneca IG, Ghiringhelli F, Zitvogel L. The intestinal microbiota modulates the anticancer immune effects of cyclophosphamide. Science. 2013 Nov 22;342(6161):971-6. doi: 10.1126/science.1240537. PMID 24264990
- [Background] Vetizou M, Pitt JM, Daillere R, Lepage P, Waldschmitt N, Flament C, Rusakiewicz S, Routy B, Roberti MP, Duong CP, Poirier-Colame V, Roux A, Becharef S, Formenti S, Golden E, Cording S, Eberl G, Schlitzer A, Ginhoux F, Mani S, Yamazaki T, Jacquelot N, Enot DP, Berard M, Nigou J, Opolon P, Eggermont A, Woerther PL, Chachaty E, Chaput N, Robert C, Mateus C, Kroemer G, Raoult D, Boneca IG, Carbonnel F, Chamaillard M, Zitvogel L. Anticancer immunotherapy by CTLA-4 blockade relies on the gut microbiota. Science. 2015 Nov 27;350(6264):1079-84. doi: 10.1126/science.aad1329. Epub 2015 Nov 5. PMID 26541610
- [Background] Sivan A, Corrales L, Hubert N, Williams JB, Aquino-Michaels K, Earley ZM, Benyamin FW, Lei YM, Jabri B, Alegre ML, Chang EB, Gajewski TF. Commensal Bifidobacterium promotes antitumor immunity and facilitates anti-PD-L1 efficacy. Science. 2015 Nov 27;350(6264):1084-9. doi: 10.1126/science.aac4255. Epub 2015 Nov 5. PMID 26541606
- [Background] Xia Y, Medeiros LJ, Young KH. Immune checkpoint blockade: Releasing the brake towards hematological malignancies. Blood Rev. 2016 May;30(3):189-200. doi: 10.1016/j.blre.2015.11.003. Epub 2015 Nov 25. PMID 26699946
- [Background] Chinai JM, Janakiram M, Chen F, Chen W, Kaplan M, Zang X. New immunotherapies targeting the PD-1 pathway. Trends Pharmacol Sci. 2015 Sep;36(9):587-95. doi: 10.1016/j.tips.2015.06.005. Epub 2015 Jul 7. PMID 26162965
- [Background] Keir ME, Butte MJ, Freeman GJ, Sharpe AH. PD-1 and its ligands in tolerance and immunity. Annu Rev Immunol. 2008;26:677-704. doi: 10.1146/annurev.immunol.26.021607.090331. PMID 18173375
- [Background] Nishimura H, Nose M, Hiai H, Minato N, Honjo T. Development of lupus-like autoimmune diseases by disruption of the PD-1 gene encoding an ITIM motif-carrying immunoreceptor. Immunity. 1999 Aug;11(2):141-51. doi: 10.1016/s1074-7613(00)80089-8. PMID 10485649
- [Background] Iwai Y, Ishida M, Tanaka Y, Okazaki T, Honjo T, Minato N. Involvement of PD-L1 on tumor cells in the escape from host immune system and tumor immunotherapy by PD-L1 blockade. Proc Natl Acad Sci U S A. 2002 Sep 17;99(19):12293-7. doi: 10.1073/pnas.192461099. Epub 2002 Sep 6. PMID 12218188
- [Background] Xu F, Xu L, Wang Q, An G, Feng G, Liu F. Clinicopathological and prognostic value of programmed death ligand-1 (PD-L1) in renal cell carcinoma: a meta-analysis. Int J Clin Exp Med. 2015 Sep 15;8(9):14595-603. eCollection 2015. PMID 26628942
- [Background] Massi D, Brusa D, Merelli B, Falcone C, Xue G, Carobbio A, Nassini R, Baroni G, Tamborini E, Cattaneo L, Audrito V, Deaglio S, Mandala M. The status of PD-L1 and tumor-infiltrating immune cells predict resistance and poor prognosis in BRAFi-treated melanoma patients harboring mutant BRAFV600. Ann Oncol. 2015 Sep;26(9):1980-1987. doi: 10.1093/annonc/mdv255. Epub 2015 Jun 2. PMID 26037795
- [Background] Brahmer JR, Drake CG, Wollner I, Powderly JD, Picus J, Sharfman WH, Stankevich E, Pons A, Salay TM, McMiller TL, Gilson MM, Wang C, Selby M, Taube JM, Anders R, Chen L, Korman AJ, Pardoll DM, Lowy I, Topalian SL. Phase I study of single-agent anti-programmed death-1 (MDX-1106) in refractory solid tumors: safety, clinical activity, pharmacodynamics, and immunologic correlates. J Clin Oncol. 2010 Jul 1;28(19):3167-75. doi: 10.1200/JCO.2009.26.7609. Epub 2010 Jun 1. PMID 20516446
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] Hodi FS, Sznol M, Kluger HM, McDermott DF, Carvajal RD, Lawrence DP. Long-term survival of ipilimumab-naive patients (pts) with advanced melanoma (MEL) treated with nivolumab (anti-PD-1, BMS-936558, ONO-4538) in a phase I trial. Journal of clinical oncology : official journal of the American Society of Clinical Oncology. 2014;32(Supplement):9002.
- [Background] McKinstry KK, Strutt TM, Swain SL. Regulation of CD4+ T-cell contraction during pathogen challenge. Immunol Rev. 2010 Jul;236:110-24. doi: 10.1111/j.1600-065X.2010.00921.x. PMID 20636812
- [Background] Ansell SM, Hurvitz SA, Koenig PA, LaPlant BR, Kabat BF, Fernando D, Habermann TM, Inwards DJ, Verma M, Yamada R, Erlichman C, Lowy I, Timmerman JM. Phase I study of ipilimumab, an anti-CTLA-4 monoclonal antibody, in patients with relapsed and refractory B-cell non-Hodgkin lymphoma. Clin Cancer Res. 2009 Oct 15;15(20):6446-53. doi: 10.1158/1078-0432.CCR-09-1339. Epub 2009 Oct 6. PMID 19808874
- [Background] Bashey A, Medina B, Corringham S, Pasek M, Carrier E, Vrooman L, Lowy I, Solomon SR, Morris LE, Holland HK, Mason JR, Alyea EP, Soiffer RJ, Ball ED. CTLA4 blockade with ipilimumab to treat relapse of malignancy after allogeneic hematopoietic cell transplantation. Blood. 2009 Feb 12;113(7):1581-8. doi: 10.1182/blood-2008-07-168468. Epub 2008 Oct 30. PMID 18974373
- [Background] Yu P, Steel JC, Zhang M, Morris JC, Waldmann TA. Simultaneous blockade of multiple immune system inhibitory checkpoints enhances antitumor activity mediated by interleukin-15 in a murine metastatic colon carcinoma model. Clin Cancer Res. 2010 Dec 15;16(24):6019-28. doi: 10.1158/1078-0432.CCR-10-1966. Epub 2010 Oct 5. PMID 20924130
- [Background] Wolchok JD, Kluger H, Callahan MK, Postow MA, Rizvi NA, Lesokhin AM, Segal NH, Ariyan CE, Gordon RA, Reed K, Burke MM, Caldwell A, Kronenberg SA, Agunwamba BU, Zhang X, Lowy I, Inzunza HD, Feely W, Horak CE, Hong Q, Korman AJ, Wigginton JM, Gupta A, Sznol M. Nivolumab plus ipilimumab in advanced melanoma. N Engl J Med. 2013 Jul 11;369(2):122-33. doi: 10.1056/NEJMoa1302369. Epub 2013 Jun 2. PMID 23724867
- [Background] Williams CD, Harrison CN, Lister TA, Norton AJ, Blystad AK, Coiffier B, Taghipour G, Schmitz N, Goldstone AH; European Bone Marrow Transplant Lymphoma Working Party. High-dose therapy and autologous stem-cell support for chemosensitive transformed low-grade follicular non-Hodgkin's lymphoma: a case-matched study from the European Bone Marrow Transplant Registry. J Clin Oncol. 2001 Feb 1;19(3):727-35. doi: 10.1200/JCO.2001.19.3.727. PMID 11157024
- [Background] Andreadis C, Schuster SJ, Chong EA, Svoboda J, Luger SM, Porter DL, Tsai DE, Nasta SD, Elstrom RL, Goldstein SC, Downs LH, Mangan PA, Cunningham KA, Hummel KA, Gimotty PA, Siegel DL, Glatstein E, Stadtmauer EA. Long-term event-free survivors after high-dose therapy and autologous stem-cell transplantation for low-grade follicular lymphoma. Bone Marrow Transplant. 2005 Dec;36(11):955-61. doi: 10.1038/sj.bmt.1705178. PMID 16205727

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: De novo diffuse large B cell lymphoma that fails to achieve a PET negative complete response to primary rituximab and anthracycline based multi-agent chemotherapy and at least maintains stable disease after salvage chemotherapy or present double/triple hit features defined by overexpression by standard immunohistochemistry of c-MYC plus BCL2 and/or BCL6 or presence of chromosomal translocations as detected by break-apart FISH involving IGH/MYC plus IGH/BCL2 and/or IGH/BCL6 and who only received standard chemoimmunotherapy with rituximab, cyclophosphamide, vincristine and prednisone (R-CHOP) for induction and present at least stable disease after consolidation or salvage chemotherapy. Stable disease (SD) for lymphoma is defined in Appendix B: Lugano Classification for Response Assessment of Non-Hodgkin Lymphoma.
- Group B: Recurrent high-risk diffuse large B cell lymphoma defined as relapsing within one year of completion of rituximab and anthracycline based multi-agent chemotherapy or a sAAIPI (second-line age-adjusted International Prognostic Index) intermediate or high at relapse or acquisition of double/triple hit features upon relapse (as defined in group A) and at least stable disease after salvage chemotherapy. Patients with an initial diagnosis of low-grade/indolent non-Hodgkin lymphoma (i.e. follicular, marginal zone) who present relapse with histologic transformation to diffuse large B cell lymphoma (confirmed by biopsy) and meet the definition for high-risk as presented above, are also eligible.
- Group C: De novo high-risk T cell lymphoma with at least stable disease after primary therapy. High risk T cell lymphoma is defined as Stage III or IV disease at presentation and/or failure to achieve CR after frontline chemotherapy. Patients with ALK-positive ALCL will be excluded from the trial. Patients with ALK-negative ALCL in complete response will be excluded from the trial.
- Group D: Recurrent T cell lymphoma with at least stable disease after salvage therapy. Patients with ALK-positive ALCL will be excluded from the trial.
- Group E: Transplant-naïve high risk multiple myeloma with at least stable disease after most recent line of therapy. High risk myeloma is defined as those carrying 1q amplifications, 1p deletions, 13q deletions by conventional cytogenetics, p53 deletions, high-risk GEP 70 scores, t(4;14), t(14;16) and t(14;20), hypodiploidy. This cohort has been discontinued due to updated risks provided by the FDA. These patients will be followed for safety and correlative studies only.
- Group F: Recurrent myeloma within 3 years after a single or tandem autologous transplant and at least stable disease after salvage therapy. Stable disease for multiple myeloma is defined in Appendix C: International Myeloma Working Group (IMWG). This cohort has been discontinued due to updated risks provided by the FDA. These patients will be followed for safety and correlative studies only.
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F
Started | 9 | 11 | 8 | 4 | 8 | 6
Completed | 6 | 6 | 6 | 4 | 6 | 4
Not Completed | 3 | 5 | 2 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Screen Failure | 2 | 4 | 2 | 0 | 1 | 1
Not completed — Discontinued Due to Updated FDA Risks | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F | Total
Number analyzed (Participants) | 9 | 11 | 8 | 4 | 8 | 6 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 5 | 5 | 3 | 0 | 5 | 27
  >=65 years | 0 | 6 | 3 | 1 | 8 | 1 | 19
Age, Continuous [Median (Full Range); unit: Years] | 51 [21 to 60] | 66 [41 to 75] | 57 [35 to 69] | 52 [26 to 72] | 69.5 [65 to 78] | 50.5 [48 to 76] | 62 [21 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 4 | 1 | 2 | 2 | 11
  Male | 8 | 10 | 4 | 3 | 6 | 4 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 2 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 0 | 3 | 5
  White | 7 | 11 | 6 | 2 | 6 | 2 | 34
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 8 | 4 | 8 | 6 | 46

OUTCOME MEASURES:

1. Primary Outcome: Safety of Combined Check Point Inhibition Therapy Via Assessment of Adverse Events and Lab Findings
Description: To assess the safety of combined check point inhibition with nivolumab and ipilimumab after autologous hematopoietic stem cell transplantation in patients at high risk for post-transplant recurrence including patients with persistent and recurrent high risk diffuse large B cell lymphoma, high risk and recurrent T cell lymphoma and high risk and recurrent multiple myeloma. The composite endpoint consisting of the occurrence of at least one treatment-related limiting toxicity (after combined checkpoint inhibitor treatment is initiated) defined as a ≥ grade 4 non-hematologic toxicity as specified by the CTCAE. If 3 of 7 patients in a single group experience a treatment-related limiting toxicity, that single group will be terminated.
Time Frame: 26 weeks
Population: Patients at high risk for post-transplant recurrence including patients with persistent and recurrent high risk diffuse large B cell lymphoma, high risk and recurrent T cell lymphoma and high risk and recurrent multiple myeloma treated with nivolumab and ipilimumab after autologous hematopoietic stem cell transplantation
Measure: Number; unit: Treatment-Related Limiting Toxicity
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F
Number analyzed (Participants) | 7 | 7 | 5 | 4 | 7 | 5
Treatment-Related Limiting Toxicity | 2 | 0 | 0 | 2 | 1 | 2

ADVERSE EVENTS:
Time Frame: From Day 1 Week 1 of combined checkpoint therapy through the end of the safety-reporting period of 100 days after the last dose of study therapy (approximately 40 weeks)
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F
All-Cause Mortality (participants affected / at risk) | 0/7 | 4/7 | 1/5 | 3/4 | 5/7 | 1/5
Serious Adverse Events (participants affected / at risk) | 3/7 | 5/7 | 2/5 | 1/4 | 4/7 | 3/5
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 5/5 | 4/4 | 7/7 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=7) | Group B (N=7) | Group C (N=5) | Group D (N=4) | Group E (N=7) | Group F (N=5)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenoviremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal Crisis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Alkaline Phosphatase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bilirubin Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-Difficile (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CPK Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
GGT Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart Block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection ESBL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
L Leg Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parainfluenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Progression Of Disease (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pseudomonas Aeruginosa Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rigors (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RSV Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis - Pseudomona Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STEMI (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
STEMI, Heart Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=7) | Group B (N=7) | Group C (N=5) | Group D (N=4) | Group E (N=7) | Group F (N=5)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Right Upper Quad) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Kidney Failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenoviremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Adrenal Insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 5 (14) | 2 (2) | 4 (8) | 1 (1) | 2 (3) | 2 (8)
Alkaline Phosphatase Increased (Investigations) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (13)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Altered Mental Status (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase Increased (Investigations) | 4 (16) | 1 (2) | 1 (1) | 2 (9) | 1 (2) | 1 (6)
Anemia (Blood and lymphatic system disorders) | 7 (18) | 6 (69) | 4 (10) | 3 (6) | 5 (31) | 4 (52)
Anemia (Intermittent) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 2 (3) | 2 (2) | 3 (5) | 1 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 5 (13) | 0 (0) | 1 (3) | 1 (1) | 2 (4) | 2 (9)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
B/L Axillary Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign Lung Tissue (Bronchoscopy Result) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bilirubin Increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (9)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blurry Vision (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blurry Vision (Intermittent) (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brachial Plexopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bump/ Mass L Occiput (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burn Right Wrist (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burning Of Back (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burning/Itching Eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-Difficile (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest Tightness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Tightness (Intermittent) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Chronic Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (7) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Constipation (Intermittent) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronavirus (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cortisol Decreased (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (9) | 2 (2) | 1 (1) | 1 (2) | 4 (4) | 1 (3)
Cough (Intermittent) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cough Sequelae Of RSV (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Cough, Dry (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CPK Increased (Investigations) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cramping Hands, Legs (Intermittent) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine Increased (Investigations) | 3 (7) | 2 (8) | 0 (0) | 0 (0) | 3 (4) | 2 (5)
Dehydration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 7 (17) | 5 (13) | 3 (11) | 2 (3) | 4 (16) | 2 (8)
Diarrhea (Intermittent) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disease Progression (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Dizziness (Intermittent) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug Reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Skin (Bl Le) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (3) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Intermittent) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Intermittent) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea On Exertion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
E.Coli In Stool (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Early Satiety (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EBV Reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Eczematous Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema (Limbs) (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema BLE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Edema LE (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema LLE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Elevated Uric Acid (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Engraftment Syndrome (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterobactercloacae In Urine (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterovirus/Rhinovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eosinophilia (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epigastric Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Burning (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Eye Burning (Intermittent) (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye Irritation L (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid Lesion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial Edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 5 (9) | 3 (5) | 3 (13) | 2 (2) | 4 (4) | 2 (6)
Fecal Urgency (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (7) | 3 (13)
Fever (Intermittent) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever/Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fevers (Intermittent) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank Pain (Right Side) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flu Like Symptoms (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Follicular Erythema Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised Pruritis (Neck, Face, Chest) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Generalized Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GGT Increased (Investigations) | 5 (10) | 1 (1) | 4 (7) | 1 (2) | 2 (2) | 3 (13)
Graft Failure/Loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haptoglobin Decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Headache (Intermittent) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hearing Impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart Failure, Systolic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heartburn (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hematuria/Dysuria/Fever (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot Flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Human Enterovirus/Rhinovirus (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Human Metapneumovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hyperglycemia Non-Fasting (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (8) | 1 (1)
Hyperglycemia Non-Fasting (Intermittent) (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperphospatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoadrenal (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypocortosolism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypogammaglobulinemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Intermittent) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3) | 4 (15) | 1 (1) | 2 (2) | 2 (4) | 2 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (6) | 2 (5) | 0 (0) | 1 (1) | 2 (5) | 2 (20)
Hypomagnesemia (Intermittent) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3) | 1 (5) | 0 (0) | 1 (1) | 2 (2) | 2 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (5) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
Hypotension (Orthostatic) (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
IGG Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune System Disorder-Hypogammaglobulinemia (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (+ Blood Culture) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection Adenovirus Reactivation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection RSV (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection Sinus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza A (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion Reaction (Sob, Feeling Cold, Rigors) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion Related (Macupapular Rash) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 2 (4)
Intermittent Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Itchy Eyes (Intermittent) (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint Pain (Intermittent) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Joint Range Of Motion Decreased (R Shoulder Rotator Cuff) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint Range Of Motion Decreased(Shoulder And Knees) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LD Increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 2 (3)
Left Arm Tingling (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left Jugular Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leg Cramps (Intermittent) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Leukocytosis (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase Increased (Investigations) | 2 (10) | 1 (2) | 1 (4) | 2 (9) | 1 (2) | 1 (7)
Localized Edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localized Edema (Left Arm) (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loose Stools (Pudding) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung Infection (Fungal Species: Mycelia Sterilia) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung Infection (Pna / Boop) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung Infection (Pna) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung Nodule (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Metapneumovirus And Coronavirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mrsa Nasal Colonization (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Mucousy Stool (Intermittent) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Left Leg) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia Bilateral Lower Extremities (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myalgias (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myopathy (Muscle Weakness Lower Limb) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myositis /Polymyalgia Secondary To Late Effects Of Ipilimumab (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 5 (10) | 1 (2) | 2 (2) | 4 (4) | 2 (5)
Nausea (Dry Heaves) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Intermittent) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathic Leg Pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Investigations) | 5 (34) | 6 (46) | 5 (23) | 2 (4) | 4 (18) | 5 (23)
Neutropenia (Intermittent) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil Count Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nodule Occipital (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Norovirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral Candidiasis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral Mucositis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Orthostatic Hypotension (Adrenal Dysfunction) (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis Media (Right) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain Calf (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain Joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain Rib (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain Right Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain Right Lower Quadrant (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain To L Flank/Rib (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain-Bl Leg Pain Chronic Back Compressed Spinal Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papular Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parainfluenza A (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parainfluenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Parainfluenza 1 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parainfluenza 3 Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paresthesia Hands (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvis Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Penile Lesion (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Peripheral Sensory Neuropathy (Intermittent) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perirectal Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phosphorous Increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postural Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pressure Ulcer (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (6) | 1 (1) | 3 (3) | 0 (0) | 3 (4) | 0 (0)
Pruritus (Intermittent) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pruritus Localised (Palm And Soles) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus Torso, Arms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Nodules (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 2 (7) | 0 (0) | 1 (1) | 1 (2)
Rash (Acneiform/Erythematous) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash (Around L Nipple) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Contact Dermatitis) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Erythematous) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Rash (Pruritic) Thighs (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Pruritic) Upper Chest (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (R Hip) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Right Hand) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash Acneiform/Erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash Erythematous (Intermittent) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash Facial (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash Hands, Back (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 2 (6) | 1 (2) | 0 (0) | 1 (1)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash Pruritic (General) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Intermittent) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash, Acneiform/Erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rashes (Macular) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rashes (Papular Lower Lid) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rashes Acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rashes Forehead (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rashes Papular (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rashes Papular Chin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Recurrent Clostridium Difficile Diarrhea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Reflux (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus/Enterovirus (Rpp Virus) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right Hip Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Right Upper Lobe Nodular Opacity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rising Blood Pressure (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shingles (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Short Term Memory Loss (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Biopsy Right Ear (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Pigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Tissue Pustules(Folliculitis) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Steroid Induced Hyperglycemia (Intermittent) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stiff Neck (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomach Discomfort/Reflux (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Investigations) | 6 (23) | 6 (32) | 3 (7) | 3 (4) | 3 (21) | 3 (40)
Thrush (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tingling Painful Hands (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremors (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremors (Hand) (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TSH Increased (Endocrine disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Burning (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Disorder Straining (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Disorder Unable To Urinate (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Enterobactercloacae Complex) (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uriticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral/Superimposed Bacterial Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (5) | 2 (3) | 0 (0) | 1 (2) | 2 (3)
Vomiting (Intermittent) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WBC Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight Loss (Investigations) | 1 (1) | 2 (18) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Wound, Sacral (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/02/NCT02681302/Prot_SAP_000.pdf